CLINICAL TRIAL: NCT07279649
Title: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis Post-Market Clinical Follow-Up (PMCF) Observational Registry
Status: Not yet recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VBX 22-08
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Aorto-iliac Occlusive Disease (AIOD); Visceral Artery Occlusive Disease (VAOD); Isolated Artery Aneurysms (IAA); Trauma or Iatrogenic Vessel Injury
Keywords: Peripheral Vascular Disease; Peripheral Arterial Disease; Aneurysm; Cardiovascular Disease; Trauma; Injury; Iliac; BXB; Aortoiliac occlusive disease; Visceral artery occlusive disease; Iliac arteries; visceral arteries; subclavian artery aneurysms; iatrogenic vessel injuries; FEVAR; BEVAR; CERAB
MeSH Terms: conditions — Wounds and Injuries; Peripheral Vascular Diseases; Peripheral Arterial Disease; Aneurysm; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Aortoiliac Occlusive Disease: De novo or rest. lesions in the iliac arteries include aortic bifurcat: Device: Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) Intent to treat with Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) in the treatment of Peripheral Artery Disease as part of routine clinical practice.
  Interventions: Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)
- Visceral Artery Occlusive Disease (VAOD): De novo or restenotic lesions in the visceral arteries: Device: Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) Intent to treat with Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) in the treatment of Peripheral Artery Disease as part of routine clinical practice.
  Interventions: Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)
- Isolated Artery Aneurysmal Disease (IAA): Isolated visceral, iliac, and subclavian artery aneurysms: Device: Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) Intent to treat with Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) in the treatment of Peripheral Artery Disease as part of routine clinical practice.
  Interventions: Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)
- Trauma or Iatrogenic Vessel Injury: are located in the chest cavity, abdominal cavity, or pelvis: Device: Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) Intent to treat with Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) in the treatment of Peripheral Artery Disease as part of routine clinical practice.
  Interventions: Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)
- Other (subjects not fitting into the categories above): Device: Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) Intent to treat with Reduced Profile GORE® VIABAHN® VBX BALLOON EXPANDABLE ENDOPROSTHESIS (BXB) in the treatment of Peripheral Artery Disease as part of routine clinical practice.
  Interventions: Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)

INTERVENTIONS:
Device: Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB) — This registry will collect data for eligible commercially available BXB device(s). The BXB device(s) will not be provided to the sites by the Sponsor. The BXB device implant procedure will be performed according to standard practice of the enrolling institution.

SUMMARY:
Collect real-world post-market clinical follow-up data on subjects treated with the Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB)

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational registry to collect real world data of the Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (Reduced Profile VBX Stent Graft-BXB) device.

The registry population will include subjects presenting with clinical conditions consistent with the BXB device indications for use and in accordance with standard of care. The following subject cohorts will be included in the registry:

* De novo or restenotic lesions in the iliac arteries including lesions at the aortic bifurcation [Aortoiliac occlusive disease (AIOD)],
* De novo or restenotic lesions in the visceral arteries [Visceral artery occlusive disease (VAOD)],
* Isolated visceral, iliac, and subclavian artery aneurysms [IAA], or
* Traumatic or iatrogenic vessel injuries in arteries that are located in the chest cavity, abdominal cavity, or pelvis (except for aorta, coronary, innominate, carotid, vertebral, and pulmonary arteries) [Arterial Injury (AI)].

To satisfy a key objective of the PMCF plan, clinical data will be collected in other indications outside of those listed above (Other cohort).

Approximately 24 clinical investigative sites in Europe, will participate in this registry. 240 subjects will be implanted in this study with a limit of 48 subjects treated / implanted per site. If a site reaches 48 subjects, enrolment will be closed for that site. All subjects will be followed through 12 months (1 year) post-procedure per standard of care. Quality of Life questionnaires will also be collected for all follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Informed Consent Form (ICF) is signed by subject
3. Suitable for endovascular treatment with the Reduced Profile GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (BXB) device
4. Willingness of the subject to adhere to institutional standard of care follow-up requirements

Exclusion Criteria:

1. Previous or concurrent enrollment into this registry (e.g., previous enrollment into another treatment cohort or subject requires enrollment into more than one cohort) (Note: Only the first treatment will be enrolled if concurrent procedures are performed that would require enrollment into more than one cohort).
2. Participation in concurrent research study or registry which may confound registry results, unless approved by Gore.
3. Known hypersensitivity to heparin, including a previous incident of Heparin-Induced Thrombocytopenia (HIT) type II.
4. Life expectancy <12 months due to comorbidities or unlikely to be available for standard of care follow-up visits as defined by sites.
5. Known intolerance to anticoagulant and / or antiplatelet therapy at the time of the index procedure
6. Subject has a known allergy to contrast or the Reduced Profile VBX Stent (BXB) device components at the time of index procedure that cannot be adequately mitigated.
7. Pregnant or breast-feeding subject at time of informed consent signature.
8. Subject has other medical conditions which, as determined by the investigator, may confound the data interpretation (e.g., sepsis, thrombophilic diseases, connective tissue disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will include subjects presenting with clinical conditions consistent with the BXB device indications for use and in accordance with standard of care. The following subject cohorts will be included in the registry:
  * Aortoiliac occlusive disease (AIOD)
  * Visceral artery occlusive disease VAOD)
  * Isolated visceral, iliac, and subclavian artery aneurysms [IAA]
  * Traumatic or iatrogenic vessel injuries in arteries that are located in the chest cavity, abdominal cavity, or pelvis (except for aorta, coronary, innominate, carotid, vertebral, and pulmonary arteries) [Arterial Injury (AI)
  * To satisfy a key objective of the PMCF plan, clinical data will be collected in other indications outside of those listed above (Other cohort) The registry has been designed with standard eligibility criteria to enroll subjects for which the registry device is intended to treat. Only subjects who meet all of the inclusion criteria and none of the exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from device-related Serious Adverse Event (SAE) for patients treated with BXB device | within 30 days after the treatment
  No adverse event that is deemed to be device-related and serious assessed by the investigator by cohort
Procedural Success for patients treated with BXB device | at the time of implant
  Successful access, delivery and deployment of BXB device, and withdrawal of catheters with patent BXB device at end of procedure

SECONDARY OUTCOMES:
Primary patency for patients treated in Aortoiliac Occlusive Disease (AIOD) through 1 year follow-up | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Blood flow through the target vessel without the need for repeat surgical or endovascular procedures
Freedom from major amputation of the BXB device treated limb for patients treated in AIOD | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  No amputation above the transmetatarsal level of the treated limb
Primary patency for patients treated in Visceral Occlusive Disease (VAOD) | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Blood flow through the target vessel without the need for repeat surgical or endovascular procedures
Survival for patients treated in VAOD | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Patient is free from death of any cause (is alive)
Freedom from reintervention through 1 year follow-up for patients treated in Isolated Artery Aneurysm (Subclavian, Visceral, Iliac) | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Freedom from unanticipated interventions on the target vessel(s) treated with the BXB Device.
30 Day Mortality for patients treated in IAA | from the time of the index procedure through 30 days
  all deaths, regardless of their relationship to the device, procedure, aneurysm, or unrelated medical conditions.
Treated vessel primary patency through 1 year follow-up for patients treated Trauma or Iatrogenic Vessel Injury | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Blood flow through the target vessel without the need for repeat surgical or endovascular procedures
Device-related adverse events (i.e. thrombosis) for patients treated in Trauma or or Iatrogenic Vessel Injury | from the time of the index procedure up to 365 days (±window, between days 335 and 455)
  Stent thrombosis deemed to be device related as assessed by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Branzan, Prof. Dr., Principal Investigator — TUM Klinikum
Locations (1):
- TUM Klinikum, Munich, Germany

IPD SHARING:
Plan to Share IPD: No